CLINICAL TRIAL: NCT03478631
Title: The Role of Dietary Nitrate on Blood Pressure and Cardiovascular Disease Risk Factors: a Randomized, Controlled Trial in Individuals With Elevated Blood Pressure
Brief Title: Dietary Nitrate on Blood Pressure and Cardiovascular Disease Risk Factors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Vladimir Vuksan, Professor, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DINO3
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Hypertension; Blood Pressure, High
Keywords: nitrate; vegetables
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, double-blind, controlled parallel study. There will be two experimental arms of 16-week duration, in which participants are assigned to test or control arms under free living conditions in an outpatient setting.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and study coordinators will be blinded to the nature of the treatment allocation. Stratified randomization lists by baseline sex and age will be created.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Nitrate Dehydrated Vegetables (Experimental): Participants are given high-nitrate dehydrated vegetable powders contained in opaque sachets. Participants are advised to consume three sachets per day, over the course of three meals, for 16 weeks.
  Interventions: Other: High-nitrate dehydrated vegetable powder
- Low-Nitrate Dehydrated Vegetables (Active Comparator): Participants are given low-nitrate dehydrated vegetable powders contained in three opaque sachets. Participants are advised to consume three sachets per day, over the course of three meals, for 16 weeks.
  Interventions: Other: Low-nitrate dehydrated vegetable powder

INTERVENTIONS:
Other: High-nitrate dehydrated vegetable powder — A mixed combination of vegetable powders that are naturally high in nitrate content, such as beet, spinach, and kale
  Arms: High Nitrate Dehydrated Vegetables
Other: Low-nitrate dehydrated vegetable powder — A mixed combination of vegetable powders that are naturally low in nitrate content, such as peas, tomato, broccoli, carrots, and brussel sprouts
  Arms: Low-Nitrate Dehydrated Vegetables

SUMMARY:
The project aims to determine the effect of a high-nitrate dietary intervention on blood pressure and markers of vascular function compared to a low-nitrate intervention in people with elevated blood pressure. Half of the participants will receive the high-nitrate dehydrated vegetable intervention, while the other half will receive the low-nitrate dehydrated vegetable intervention.This project will advance the current hypothesis on the therapeutic link between dietary nitrate and high blood pressure, and potentially derive impactful recommendations for individuals at risk of hypertension.

DETAILED DESCRIPTION:
Diets rich in fruits and in particular, vegetables, reduce blood pressure (BP) and the risk of cardiovascular events. Increasingly, attention is being given to high-nitrate containing vegetables, with emerging evidence that it might represent a source of vasoactive nitric oxide. Clinical data to date uniformly suggest an acute vasoprotective role of dietary nitrate administration and a BP-lowering effect. Whether the vascular effects extend to long-term intake and in individuals with elevated blood pressure is not well known. The investigators hypothesize that consumption of a dietary intervention high in nitrate from vegetable sources will have a greater effect on BP and related vascular parameters than a similar intervention that is low in dietary nitrates.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-35 kg/m2
* Seated systolic blood pressure ≥130 and <160 mmHg

Exclusion Criteria:

* current use of antihypertensive agents
* history of major cardiovascular events in the last 1 year (stroke or myocardial infarction)
* stage II hypertension as per JNC7 criteria (systolic BP/ diastolic BP ≥160/100 mmHg) - angina pectoris
* gastrointestinal (i.e. inflammatory bowel disease, celiac), liver or kidney disease
* cardiac condition that compromises normal function (e.g. mitral valve disease, heart failure)
* serum triglyceride >4.5mmol/L
* major disability or disorder requiring continuous medical attention
* planned initiation in antihypertensive therapy
* herb or supplement use that may affect primary outcome
* consuming >3 servings of vegetables/day (based on semi-quantitative food frequency questionnaire)
* alcohol use >2 drinks/day
* chronic or prescribed use of medications including prescription NSAIDs, antacids, warfarin, medications affecting NO synthesis (ie. sildenafil, organic nitrates, etc)
* use of antibiotics within 3-months of the study start
* participants should also be willing to refrain from using mouthwash (ie chlorhexidine) for the duration of their participation in the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Baseline, 8 and16 weeks
  Change in systolic blood pressure vs. control at 16 weeks

SECONDARY OUTCOMES:
Mean 24h and Daytime Ambulatory Systolic, Diastolic and Mean Arterial Blood Pressure | Baseline and 16 weeks
  Change in mean 24h and daytime ambulatory systolic, diastolic and mean arterial blood pressure vs. control at 16 weeks
Aortic Systolic and Diastolic Blood Pressure | Baseline, 8 and 16 weeks
  Change in aortic systolic and diastolic blood pressure vs. control at 16 weeks
Pulse Wave Velocity (PWV) | Baseline and 16 weeks
  Change in PWV vs. control at 16 weeks
Augmentation Index (AI) | Baseline, 8 and 16 weeks
  Change in AI vs. control at 16 weeks
High Sensitivity C-reactive protein (hs-CRP) | Baseline and 16 weeks
  Change in hs-CRP vs. control at 16 weeks
Plasma Lipids | Baseline and 16 weeks
  Change in Total-C, LDL-C, HDL-C vs. control at 16 weeks

OTHER OUTCOMES:
Symptoms Diary | Screening, baseline, 8 and 16 weeks
  Record of any adverse symptoms experienced and the level of severity
Aspartate Aminotransferase (AST) | Screening, baseline, 8 and 16 weeks
  Liver function test
Creatinine | Screening, baseline, 8 and 16 weeks
  Kidney function test
Sachet Count | 8 and 16 weeks
  Record of the amount of sachets and contents returned
7-Day Food Record | Baseline, 8 and 16 weeks
  Record of food intake 7 days prior to study visit day
Nitrate Food Frequency Questionnaire | Biweekly (screening, 0,2,4,6,8,10,12,14,16,18 weeks)
  Assess consumption of nitrate-rich meats and vegetables
Habitual Physical Activity Questionnaire | Baseline, Week 16
  Questions to assess level of physical activity
Body Weight | Screening, baseline, 8 and 16 weeks
  Body Weight in kg
24h Urinary Nitrite and Nitrate levels (exploratory outcome, TBD) | 16 weeks
  Marker of treatment compliance
24h Urinary Potassium levels (exploratory outcome, TBD) | 16 weeks
  Urine samples collected for estimation of potassium intake
24h Urinary Sodium levels (exploratory outcome, TBD) | 16 weeks
  Urine samples collected for estimation of sodium intake
Cyclic guanosine monophosphate (cGMP) (exploratory outcome, TBD) | Baseline and 16 weeks
  Change in cGMP vs. control at 16 weeks
Plasma nitrate/nitrite (exploratory outcome, TBD) | Baseline and 16 weeks
  Change in plasma nitrate and nitrite vs. control at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No